CLINICAL TRIAL: NCT02289495
Title: A Double Blind, Placebo Controlled, Single and Repeat Dose Escalation Study of GSK2838232 With and Without Ritonavir for 8-11 Days in Healthy Subjects
Brief Title: A Repeat Dose Pharmacokinetic (PK) and Safety Study of GSK2838232 With and Without Ritonavir (RTV) Conducted in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200207
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Single Dose Escalation; Repeat Dose Escalation; GSK2838232; Ritonavir
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — GSK-2838232; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2838232 without RTV (Experimental): Subjects will receive 20 mg of GSK2838232/ placebo (3:1) in cohort 1 and 50 mg of GSK2838232/ placebo (3:1) in cohort 2, administered QD for 8 days. There will be a minimum period of 7 days between successive cohorts to establish safety and PK for dose escalation; enrollment into a cohort will commence following review of interim PK and safety data from at least 4 subjects in the preceding cohort
  Interventions: Drug: GSK2838232; Drug: Placebo
- GSK2838232 with RTV (Experimental): Subjects will receive 10 mg of GSK2838232/ placebo (3:1) in cohort 3, 20 mg of GSK2838232/ placebo (3:1) in cohort 4 and 50 mg of GSK2838232/ placebo (3:1) in cohort 5, co administered with RTV 100 mg, QD for 11 days. There will be a minimum period of 7 days between successive cohorts to establish safety and PK for dose escalation; enrollment into a cohort will commence following review of interim PK and safety data from at least 4 subjects in the preceding cohort
  Interventions: Drug: GSK2838232; Drug: Placebo; Drug: Ritonavir

INTERVENTIONS:
Drug: GSK2838232 — GSK2838232 will be available as oral suspension dispersion in hydromellulose acetate succinate bulk powder/10, 20 and 50 mg which is to be administered orally QD for 8 days (Part A) or 11 days (Part B), morning dose, following an overnight fast of at least 10 hours
Drug: Placebo — Matching placebo of Suspension to active dose, administered orally QD for 8 days (Part A) or 11 days (Part B), morning dose, following an overnight fast of at least 10 hours
Drug: Ritonavir — Ritonavir will be available as white film-coated ovaloid tablets of 100 mg tablet/100mg to be administer orally, QD
  Arms: GSK2838232 with RTV

SUMMARY:
The proposed study, 200207 is a double blind, placebo controlled, single and repeat dose escalation study to investigate the safety, tolerability and PK of GSK2838232 alone and when co-administered with RTV 100 milligram (mg) Once daily (QD). This study will enable future clinical development of GSK2838232 in healthy subjects and in a Phase IIa proof of concept study in Human Immunodeficiency Virus (HIV) infected patients. This study is a single and repeat dose escalation study and will be conducted as two Parts. Part A will evaluate GSK2838232 20 mg and 50 mg administered QD for 8 days and Part B will evaluate GSK2838232 10 mg, 20 mg, and 50 mg, co-administered with RTV 100 mg, QD for 11 days. The extended period of dosing is to account for the longer terminal phase half-life of GSK2838232 when given with RTV. Dose cohorts will be enrolled sequentially; enrollment into a cohort will commence following review of interim PK and safety data from at least 4 subjects in the preceding cohort. Subjects in both parts will have a screening visit within 30 days prior to first dose and a follow-up visit 7-14 days after the last dose. Maximum duration of study participation will be approximately 7 weeks. Approximately 40 healthy subjects will be enrolled, 8 subjects/cohort. Subjects will be randomized 3:1 to receive GSK2838232 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A Creatinine clearance (CLcr) >80 millilitre per minute (mL/min) as determined by Cockcroft-Gault equation where age is in years, weight (Wt) is in kg, and serum creatinine (Scr) is in units of milligram / decilitre (mg/dL); CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (times 0.85 if female).
* Body weight >= 50 kilogram (kg [110 pounds {lbs}]) for men and >= 45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kilogram per meter square kg/m^2 (inclusive)
* Male or Female; Female subject of non-reproductive potential : is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until one week after the last dose of study medication. a) Vasectomy with documentation of azoospermia, b) Male condom plus partner use of one of the contraceptive options below: Contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label, Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label, Oral Contraceptive, either combined or progestogen alone Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects who have asthma or a history of asthma.
* Medical history of cardiac arrhythmias or cardiac disease or a family and personal history of long QT syndrome.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* Screening or baseline cardiac troponin I greater than the 99% cutoff (>.045 nanogram/ milliliter [ng/mL] by the Dimension Vista Cardiac troponin assay).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Exclusion Criteria for 24-Hour Screening Holter: Any symptomatic arrhythmia (except isolated extra systoles), Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, supraventricular tachycardia (>=10 consecutive beats), complete heart block). Non-sustained or sustained ventricular tachycardia (defined as >= 3 consecutive ventricular ectopic beats). Any conduction abnormality (including but not specific to left or right incomplete or complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolff-Parkinson-White [WPW] syndrome etc.). Sinus Pauses > 3 seconds. 300 or more supraventricular ectopic beats in 24 hours. 250 or more ventricular ectopic beats in 24 hours.
* Any clinically significant abnormal echocardiogram finding. Abnormal echocardiogram findings should be discussed with the Medical Monitor prior to enrolment.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate <45 and >100 beats per minute (bpm) (Males); <50 and >100 bpm (Males); For both Males and Females: PR Interval <120 and >220 msec, QRS duration <70 and >120 millisecond (msec); QTc interval (Fridericia's) >450 msec. Notes: A heart rate from 100 to 110 bpm can be rechecked by ECG or vitals within 30 minutes to verify eligibility. Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization). Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], WPW syndrome). Sinus Pauses > 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator or GlaxoSmithKline medical monitor, will interfere with the safety for the individual subject. Non-sustained or sustained ventricular tachycardia (>= 3 consecutive ventricular ectopic beats).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2015-06-27 (Actual); Study Completion 2015-06-27 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) assessments | Up to approximately 7 weeks
  Safety was assessed by monitoring AE and serious AEs (SAE). AEs and SAEs will be collected from the start of Study Treatment until the follow-up contact
Safety assessed by laboratory evaluations | Up to approximately 7 weeks
  Laboratory evaluations will include hematology, clinical chemistry, urinalysis assessments
Vital signs assessments | Up to approximately 7 weeks
  Vital signs will be measured in semi-supine position after 10 minutes rest and will include systolic and diastolic blood pressure and pulse rate.
Electrocardiogram (ECG) parameters assessments | Up to approximately 7 weeks
  Triplicate OR Single 12-lead ECGs will be obtained at each timepoint during the study after a 10 minute rest using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Composite pharmacokinetic profile of GSK2838232, , with and without RTV for Part A and Part B | Up to 144 hours post dose of Day 11
  PK assessments will include: On Day 1: Area under the concentration-time curve over the dosing interval (AUC[0 tau], Maximum observed concentration (Cmax), Pre-dose (trough) concentration at the end of the dosing interval (Ctau), time of occurrence of Cmax (tmax), lag time before observation of drug concentrations in sampled matrix (tlag), on Day 8 (Part A) or Day 11 (Part B): AUC(0-tau), Cmax, Ctau, tmax, tlag, terminal phase half-life (t1/2), last observed quantifiable concentration (Clast), time of last quantifiable concentration (tlast), Apparent clearance following oral dosing (CL/F).

SECONDARY OUTCOMES:
Composite pharmacokinetic profile of GSK2838232 to dose proportionality with and without RTV | Up to Day 17
  GSK2838232 AUC(0-tau), Cmax, Ctau
Composite pharmacokinetic profile to assess accumulation of GSK2838232 with and without RTV | Up to Day 17
  Accumulation will also be evaluated for each treatment by determining the ratio of Day 8 (Part A) or Day 11 (Part B) to Day 1 AUC(0 tau) (ratio of [AUC{0-tau}]), Cmax (R[Cmax]), and Ctau (R[Ctau])
Pharmacokinetic profile to assess time to steady-state of GSK2838232 with and without RTV | Up to Day 17
  Pre-dose concentrations on Day 2-8 (Part A) and Day 2-11 (Part B)
Pharmacokinetic profile to compare the pharmacokinetics of GSK2383232 with and without RTV | Up to Day 17
  GSK2838232 AUC(0-tau), Cmax, and Ctau

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- See also: Results for study 200207 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200207?search=study&b'search_terms=200207'#rs